CLINICAL TRIAL: NCT00455702
Title: Effects of Weekly Dosing of D-cycloserine on Cognitive Function in Individuals
Brief Title: Effects of Weekly Dosing of D-cycloserine on Cognitive Function in Individuals With Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Donald C. Goff, MD, Director of the Schizophrenia Clinical and Research Program, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2005-P-001040
Record Dates: First submitted 2007-04-02; First posted 2007-04-04 (Estimated); Results first posted 2014-08-07 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-07

CONDITIONS: Schizophrenia
Keywords: schizophrenia; cognition; d-cycloserine; memory
MeSH Terms: conditions — Schizophrenia | interventions — Cycloserine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- D-cycloserine (Experimental): 50 mg d-cycloserine
  Interventions: Drug: d-cycloserine
- Placebo (Placebo Comparator): 50 mg placebo
  Interventions: Drug: d-cycloserine

INTERVENTIONS:
Drug: d-cycloserine — 50mg dose d-cycloserine v placebo

SUMMARY:
The study aims to assess the effects of single dose and repeated weekly dosing of 50mg d-cycloserine versus placebo on cognitive and memory functioning in schizophrenia patients. The study will also examine the effects of 50mg d-cycloserine on positive symptoms and negative symptoms, as well as assess tolerability and side-effects.

DETAILED DESCRIPTION:
This is a ten-week, parallel-group, placebo-controlled trial examining the cognitive effects at weeks 1, 2, 3. 4, 5, 6, 7, 8 & 10 of once-weekly oral D-cycloserine 50 mg added to a stable dose of antipsychotic for 8 weeks in 60 adult outpatients with schizophrenia.

Specific aims:

1. Assess the effects of a single dose of D-cycloserine 50 mg on cognitive functioning compared to placebo.
2. Assess the effects of repeated weekly dosing of D-cycloserine on cognitive functioning at week 8 compared to placebo.
3. Assess the effects of repeated weekly dosing of D-cycloserine on memory functioning once a week 1 hour after medication administration compared to placebo.
4. Assess the persistence of learned information in a no-treatment follow-up assessment at Week 10 in the D-cycloserine group compared to the placebo group.
5. Assess effects of weekly D-cycloserine dosing on positive & negative symptoms at week 8 compared to placebo.
6. Assess tolerability and side effects of weekly D-cycloserine compared to placebo.
7. Assess the effects of d-cycloserine dosed weekly for seven weeks on reward responsiveness as measured with the response bias task compared with placebo.
8. Assess the effects of d-cycloserine dosed weekly for seven weeks on measures of functioning.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. Age 18-65 years
3. Diagnosis of schizophrenia or schizoaffective disorder, depressed type
4. Stable dose of antipsychotic for at least 4 weeks.
5. Able to provide informed consent
6. Able to complete a cognitive battery

Exclusion Criteria:

1. Current treatment with clozapine
2. Dementia
3. Seizure disorder
4. Unstable medical illness
5. Active substance abuse
6. Pregnancy, nursing, or unwilling to use appropriate birth control measures during participation if female and fertile.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2004-07; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald C Goff, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Goff DC, Cather C, Gottlieb JD, Evins AE, Walsh J, Raeke L, Otto MW, Schoenfeld D, Green MF. Once-weekly D-cycloserine effects on negative symptoms and cognition in schizophrenia: an exploratory study. Schizophr Res. 2008 Dec;106(2-3):320-7. doi: 10.1016/j.schres.2008.08.012. Epub 2008 Sep 16. PMID 18799288

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were stable adult outpatients at an urban community mental health center, ages 18-65 years, with a diagnosis of schizophrenia .
Period: Overall Study
Arm/Group | D-cycloserine | Placebo
Started | 19 | 19
Completed | 16 | 16
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | D-cycloserine | Placebo | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 19 | 38
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (9.15) | 48 (6.66) | 49.05 (7.905)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 10 | 13 | 23
Region of Enrollment [Number; unit: participants]
  United States | 19 | 19 | 38

OUTCOME MEASURES:

1. Primary Outcome: Main Outcome Measure: The Change From Baseline to Week 8 on the SANS
Description: The change from baseline to week 8 on the scale for the assessment of negative symptoms (SANS) total score. Total SANS scores range from 0-100. The SANS is comprised of 5 subscores: Affective Flattening or Blunting (score range 0-35), Alogia (score range 0-20), Avolition-Apathy (score range 0-15), Anhedonia-Asociality (score range 0-20), and Attention (0-10). For each scale, the higher the score the more prominent the negative symptoms were. The total score was computed by adding all the subscale total scores. To compute change in scores, week 8 scores were subtracted from baseline scores, resulting in a change score. Higher values equals greater improvement (i.e. week 8 score was lower than baseline score).
Time Frame: Baseline score vs. Week 8
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | D-cycloserine | Placebo
Number analyzed (Participants) | 16 | 17
Units on a scale | 2.06 (5.03) | -2.11 (7.05)

2. Secondary Outcome: Treatment Effects on the Positive Syndrome Subscale of the PANSS
Description: The change from baseline to week 8 on the positive symptom sub-scale of the Positive and Negative Syndrome Scale (PANSS). Total PANSS positive symptom sub-scale scores range from 7-49. The PANSS positive symptom sub-scale is comprised of 7 items rated on a scale of 1-7: delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, and hostility. A score of one on each item 1 absent, 2 is minimal, 3 is mild, 4 is moderate, 5 is moderately severe, 6 is severe, and 7 is extreme. The total score was computed by adding all the items on the sub-scale together. To compute change in scores, week 8 scores were subtracted from baseline scores, resulting in a change score. Higher values equals greater improvement (i.e. week 8 score was lower than baseline score).
Time Frame: Baseline score vs. Week 8 score
Population: One participant from the placebo group was removed from this analysis.
Measure: Mean (Standard Deviation); unit: PANSS Positive Subscale Units
Arm/Group | D-cycloserine | Placebo
Number analyzed (Participants) | 16 | 16
PANSS Positive Subscale Units | .19 (2.10) | -.19 (4.65)

ADVERSE EVENTS:
Arm/Group | D-cycloserine | Placebo
Serious Adverse Events (participants affected / at risk) | 1/19 | 0/19
Other Adverse Events (participants affected / at risk) | 8/19 | 13/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | D-cycloserine (N=19) | Placebo (N=19)
Worsening psychosis due to discontinuation of anti-psychotic (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | D-cycloserine (N=19) | Placebo (N=19)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Anxiety (Social circumstances) | 0 (0) | 1 (1)
Chest pain (Cardiac disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 1 (1) | 0 (0)
Fracture (foot) (General disorders) | 0 (0) | 1 (1)
Headache (General disorders) | 2 (2) | 0 (0)
Nausea (General disorders) | 0 (0) | 1 (1)
URI (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Vertigo (General disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Heartburn (Gastrointestinal disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
As the first study of once-weekly dosing in Schizophrenia, this study was exploratory and so results must be considered preliminary. Additional studies are needed to replicate these findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No